CLINICAL TRIAL: NCT00508482
Title: A Clinical Standardization Study of the Preferred Acupuncture Treatment Protocol to Treat Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Zhishun, Chief of the Acupuncture Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006BAI12B05-1
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Constipation
Keywords: Acupuncture; Functional constipation
MeSH Terms: conditions — Constipation | interventions — Acupuncture Therapy; Electroacupuncture; Lactulose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- deep needling group (Experimental): Acupoints of bilateral Tianshu (ST25), which were located according to WHO Standardized Acupuncture Points Location, were used. After sterilizing the skin, needles of the size of 0.35×0.75mm were inserted into ST25 vertically and slowly without manipulation for about 20~60mm until piercing into the muscle layer. Paired alligator clips of the electric acupuncture (EA) apparatus were attached transversely to the needle holders of bilateral ST25. EA stimulation lasted for 30 minutes with a dilatational wave of 2/15Hz and current intensity of 0.1~1mA. Participant's abdominal muscle twitching mildly showed the proper dose. Patients were treated once a day, five times a week for continuous 4 weeks.
  Interventions: Other: deep needling
- lactulose group (Active Comparator): Lactulose Oral Solution was taken orally at the dose of 20~30ml once every morning after breakfast for continuous 4 weeks. Patients should take lactulose for another 3 months if no severe adverse effect was showed.
  Interventions: Drug: Lactulose
- shallow needling group (Active Comparator): Bilateral ST25, the same acupoints as deep needling group, were used. After skin disinfection, needles of the size of 0.30×25mm penetrated the skin uprightly for about 5~9mm into the fat layer without manipulation. The usage of EA apparatus and treatment course were the same as deep needling group.
  Interventions: Other: shallow needling

INTERVENTIONS:
Other: deep needling — Huatuo brand needle (0.35×75mm), LH202H electric stimulator, parameter is constant wave, 2/15Hz, and current intensity is the abdominal muscles shiver slightly and the patient feels trivial pain.
  Once a day, five times a week, four weeks.
  Other Names: acupuncture; electroacupuncture
  Arms: deep needling group
Drug: Lactulose — 20-30ml, once a day before breakfast, for the whole study except the run-in period
  Other Names: Lactulose produced by Solvay Pharmaceuticals BV
  Arms: lactulose group
Other: shallow needling — Huatuo brand needle (0.30×25mm). The usage of EA apparatus and treatment course were the same as deep needling group.
  Other Names: acupuncture; electroacupuncture
  Arms: shallow needling group

SUMMARY:
The purpose of this study is to re-evaluate the therapeutic superiority and safety of acupuncture treatment using high quality and large sampled clinical research. The investigators want to provide a preferred treatment protocol, which is effective, safe, and easy to use in clinical practice. This research also clarifies that the insertion depth is a key factor in the therapeutic effect of acupuncture. The results of the study will help promote the development of the standardization of acupuncture.

DETAILED DESCRIPTION:
Functional constipation is a high morbidity disease. The life-long treatment of functional constipation can seriously impact a patient's quality of life. At present, one of the most frequently used treatment is catharsis, which deals with the symptom. There are three main problems with catharsis. First, there are no long-lasting effects once the patient stops taking medication. Second, there are many side effects, including abdominal pain with defecation and diarrhea. Third, long-term use of irritant laxatives will not only make the constipation become refractory and complex; but also, this type of medicine can harm the enteric nervous system, cause melanosis coli, or even carcinoma of colon. Therefore, a therapy that is safe with minimal side effects and good short-term and long-term effects is urgently needed in functional constipation treatment.

Clinical practice shows that acupuncture may meets this need to some extent. The acupuncture therapy is safe and effective and the therapeutic effects are still present several months after the treatment has been completed.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnosis of Rome III criteria;
* aged from 18 to 75 years old;
* no use of medicine for constipation about 2 weeks before the enrollment, no acupuncture treatment for constipation in the previous 3 months, and never joined any other trial in progress in the previous 3 months;
* volunteered to join this trial and signed the informed consent form

Exclusion Criteria:

* irritable bowel syndrome, organic constipation or secondary constipation caused by endocrine, metabolic, nervous, postoperative diseases, or by drugs;
* constipation with serious cardiovascular, hepatic or renal diseases, cognitive dysfunction, aphasia, mental disorders, or illness which affects the cooperation for examination and treatment;
* women in gestation or lactation period;
* abdominal aortic aneurysm or hepatosplenomegaly, etc.;
* blood coagulation disorders or using anticoagulants regularly such as Warfarin and Heparin;
* cardiac pacemaker carrier.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, M.D., Study Director — Guang'an Men Hospital Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospital Affiliated to China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wu J, Liu B, Li N, Sun J, Wang L, Wang L, Cai Y, Ye Y, Liu J, Wang Y, Liu Z. Effect and safety of deep needling and shallow needling for functional constipation: a multicenter, randomized controlled trial. Medicine (Baltimore). 2014 Dec;93(28):e284. doi: 10.1097/MD.0000000000000284. PMID 25526462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ot this trial started in April 2008 and finished in Dec. 2010. Patients were recruited from clinics in each center by posters and advertisements in newspapers.
Groups:
- Deep Needling Group: Acupoints of bilateral Tianshu (ST25), which were located according to WHO Standardized Acupuncture Points Location20, were used.
  After sterilizing the skin, needles of the size of 0.35×0.75mm were inserted into ST25 vertically and slowly without manipulation for about 30~70mm until touching the parietal peritoneum. Paired alligator clips of the EA apparatus were attached transversely to the needle holders of bilateral ST25. EA stimulation lasted for 30 minutes with a dilatational wave of 2/15Hz and current intensity of 0.1~1mA. Participant's abdominal muscle twitching mildly showed the proper dose.
  Patients were treated once a day, five times a week for continuous 4 weeks.
Period: Over 4 Weeks of Treatment
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Started | 237 | 119 | 119
Completed | 216 | 102 | 99
Not Completed | 21 | 17 | 20
Not completed — Changed mind, didn't want to participate | 9 | 7 | 4
Not completed — Lost to Follow-up | 12 | 10 | 16
Period: at the 4th Week of Follow-up
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Started | 216 | 102 | 99
Completed | 196 | 96 | 98
Not Completed | 20 | 6 | 1
Not completed — Lost to Follow-up | 20 | 6 | 1
Period: at the 12th Week of Follow-up
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Started | 196 | 96 | 98
Completed | 196 | 96 | 98
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group | Total
Number analyzed (Participants) | 237 | 119 | 119 | 475
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 0 | 4
  Between 18 and 65 years | 199 | 101 | 101 | 401
  >=65 years | 35 | 17 | 18 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.18 (17.28) | 45.21 (17.40) | 43.71 (17.23) | 44.87 (17.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 91 | 98 | 372
  Male | 54 | 28 | 21 | 103
Race/Ethnicity, Customized [Number; unit: participants]
  Han | 229 | 115 | 114 | 458
  Minority | 8 | 4 | 5 | 17
Region of Enrollment [Number; unit: participants]
  China | 237 | 119 | 119 | 475
mean spontaneous bowel movements [Median (Inter-Quartile Range); unit: stools/week] — defecation times in one week without help of medication or hands
  stools/week | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
straining during defecation [Median (Inter-Quartile Range); unit: units on a scale] — one of symptoms assessed by patients (including four symptoms) at baseline.It ranges from 0 to 4. '0' means no such symptom and '4' means very severe symptom.
  units on a scale | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3]
Incomplete evacuation [Median (Inter-Quartile Range); unit: units on a scale] — one of symptoms assessed by patients (including four symptoms) at baseline. It ranges from 0 to 4. '0' means no such symptom and '4' means very severe symptom.
  units on a scale | 2 [2 to 3] | 2 [2 to 3] | 2 [1 to 3] | 2 [2 to 3]
Stool consistency [Median (Inter-Quartile Range); unit: units on a scale] — one of symptoms assessed by patients (including four symptoms) at baseline. It ranges from 0 to 4,among them '0' means normal faeces and '4' means very hard faeces.
  units on a scale | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3]
abdominal distention [Median (Inter-Quartile Range); unit: units on a scale] — one of symptoms assessed by patients (including four symptoms) at baseline. It ranges from 0 to 4. '0' means no such symptom and '4' means very severe symptom.
  units on a scale | 1 [1 to 2] | 2 [1 to 2] | 1 [0 to 2] | 1 [0 to 2]
Cleveland Clinic Score [Median (Inter-Quartile Range); unit: units on a scale] — A scale about constipation symptoms, assessed by the doctor. There are eight items(the score was summed up by the 8 items). It ranges from '0' to '30'. '0' means none of symptoms and '30' means very severe symptoms.
  units on a scale | 13 [11 to 16] | 13 [11 to 16] | 13 [10 to 15] | 13 [10 to 15.25]

OUTCOME MEASURES:

1. Primary Outcome: Change of Mean Weekly Spontaneous Bowel Movements
Description: Spontaneous bowel movements per week were assessed every week during 4 weeks of treatment according to patients' diaries. Weekly spontaneous bowel movements were also assessed at the 4th and 12th week of follow-up according to patients' diaries.
Time Frame: over 4-week treatment, at the 4th week of follow-up, at the 12th week of follow-up
Population: Intention-To-Treat(ITT) analysis was used.
Measure: Median (Inter-Quartile Range); unit: stools/week
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
stools/week
  over 4 weeks of treatment | 2 [1.25 to 3] | 2 [1 to 2.75] | 2 [1 to 3]
  at the 4th week of follow-up | 2 [1 to 3] | 2 [0 to 3] | 1 [0 to 2]
  at the 12th week of follow-up | 2 [0.5 to 3] | 1.5 [0.5 to 3] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Comparison among three groups over 4 weeks of treatment; Test type: Superiority or Other; p = 0.238, Kruskal-Wallis
Statistical Analysis 2: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Comparison among three groups at the 4th week of follow-up; Test type: Superiority or Other; p = 0.004, Kruskal-Wallis
Statistical Analysis 3: Comparison: Deep Needling Group vs Shallow Needling Group; at the 4th week of follow-up; Test type: Superiority or Other; p = 0.277, Least-Significant Difference; We translated the data of three groups through rank cases, so that we can use Least-Significant Difference for the comparison of any two groups
Statistical Analysis 4: Comparison: Deep Needling Group vs Lactulose Group; at the 4th week of follow-up; Test type: Superiority or Other; p = 0.001, Least-Significant Difference; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 5: Comparison: Shallow Needling Group vs Lactulose Group; at the 4th week of follow-up; Test type: Superiority or Other; p = 0.055, Least-Significant Difference; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 6: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Comparison among three groups at the 12th week of follow-up; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis
Statistical Analysis 7: Comparison: Deep Needling Group vs Shallow Needling Group; at the 12th week of follow-up; Test type: Superiority or Other; p = 0.330, Least-Significant Difference; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 8: Comparison: Deep Needling Group vs Lactulose Group; at the 12th week of follow-up; Test type: Superiority or Other; p < 0.001, Least-Significant Difference; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 9: Comparison: Shallow Needling Group vs Lactulose Group; at the 12th week of follow-up; Test type: Superiority or Other; p = 0.018, Least-Significant Difference; [statistical method as in outcome 1, analysis 3]

2. Secondary Outcome: Change of Mean Value of Straining During Defecating
Description: Score of straining during defecating was assessed every week according to patients' diaries during 4 weeks of treatment. Score ranges from '0' to '4'. '0' means none of symptoms and '4' means very severe symptoms. Change from baseline of the mean value of straining during defecating over 4 weeks of treatment was evaluated as the secondary outcome. The change was calculated as the value at baseline minus the average over 4 weeks of treatment. We corrected the mean value of straining during defecating by covariance because the data had significant difference among three groups at baseline.
Time Frame: over 4 weeks of treatment
Population: ITT analysis was used
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
units on a scale | 0.835 (0.037) [0.25 to 1.5] | 0.789 (0.053) [0.06 to 1.5] | 0.868 (0.053) [0 to 1.5]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.573, ANOVA

3. Secondary Outcome: Change of Mean Value of Incomplete Evacuation
Description: Score of incomplete evacuation was assessed every week according to patients' diaries during 4 weeks of treatment. Score ranges from '0' to '4'. '0' means none of symptoms and '4' means very severe symptoms. Change from baseline of the mean value of incomplete evacuation over 4 weeks of treatment was evaluated as the secondary outcome. The change was calculated as the value at baseline minus the average over 4 weeks of treatment.
Time Frame: over 4 weeks of treatment
Population: ITT analysis was used.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
units on a scale | 0.75 [0 to 1.5] | 0.75 [0 to 1.5] | 0.75 [-0.25 to 1.25]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.271, Kruskal-Wallis

4. Secondary Outcome: Change of Mean Value of Stool Consistency
Description: Score of stool consistency was assessed every week according to patients' diaries during 4 weeks of treatment. Score ranges from '0' to '4'. '0' means none of symptoms and '4' means very severe symptoms. Change from baseline of the mean value of stool consistency over 4 weeks of treatment was evaluated as the secondary outcome. The change was calculated as the value at baseline minus the average over 4 weeks of treatment. We corrected the mean value of stool consistency by covariance because the data had significant difference among three groups at baseline.
Time Frame: over 4 weeks of treatment
Population: ITT analysis was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
units on a scale | 0.414 (0.025) [0 to 1] | 0.438 (0.035) [0 to 1] | 0.701 (0.035) [0 to 1]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Deep Needling Group vs Shallow Needling Group; Test type: Superiority or Other; p = 0.580, Least-Significant Difference
Statistical Analysis 3: Comparison: Deep Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Least-Significant Difference
Statistical Analysis 4: Comparison: Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Least-Significant Difference

5. Secondary Outcome: Change of Mean Value of Abdominal Distention
Description: Score of abdominal distention was assessed every week according to patients' diaries during 4 weeks of treatment. Score ranges from '0' to '4'. '0' means none of symptoms and '4' means very severe symptoms. Change from baseline of the mean value of abdominal distention over 4 weeks of treatment was evaluated as the secondary outcome. The change was calculated as the value at baseline minus the average over 4 weeks of treatment. We corrected the mean value of abdominal distention by covariance because the data had significant difference among three groups at baseline.
Time Frame: over 4 weeks of treatment
Population: ITT analysis was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Shallow Needling Group: Bilateral ST25, the same acupoints as deep needling group, were used. After skin disinfection, needles of the size of 0.30×25mm penetrated the skin uprightly for about 5~9mm into the fat layer without manipulation. The usage of EA apparatus and treatment course were the same as deep needling group.
  .
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
units on a scale | 0.762 (0.033) [5 to 9] | 0.693 (0.041) [6 to 9] | 0.661 (0.047) [6 to 11]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.167, ANOVA

6. Secondary Outcome: Change of Mean Value of Cleveland Clinic Score
Description: Cleveland Clinic Score was assessed by doctors which contains eight items about constipation-related symptoms. Score ranges from '0' to '30'. '0' means none of symptoms and '30' means very severe symptoms. The change was calculated as the value at baseline minus the average over 4 weeks of treatment.
Time Frame: over 4 weeks of treatment
Population: ITT analysis was used
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
units on a scale | 4.5 [2.25 to 7.25] | 4.38 [1.06 to 6.44] | 4 [1.25 to 6.25]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.066, Kruskal-Wallis

7. Secondary Outcome: Time to the First Spontaneous Bowel Movement After the First Treatment
Time Frame: counting by hours
Population: ITT analysis was used
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
hours | 27.08 (27.53) [2 to 3] | 36.68 (32.75) [2 to 3] | 16.52 (18.84) [2 to 2]
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Deep Needling Group vs Shallow Needling Group; Test type: Superiority or Other; p = 0.024, Least-Significant Difference
Statistical Analysis 3: Comparison: Deep Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Least-Significant Difference
Statistical Analysis 4: Comparison: Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Least-Significant Difference

8. Secondary Outcome: Percentage of the Usage of Emergency Drugs
Time Frame: over 4 weeks of treatment
Population: ITT analysis was used.
Measure: Number; unit: percentage of participants
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
percentage of participants | 9.65 | 8.04 | 33.91
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Deep Needling Group vs Shallow Needling Group; Test type: Superiority or Other; p = 0.627, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)
Statistical Analysis 3: Comparison: Deep Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)
Statistical Analysis 4: Comparison: Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)

9. Secondary Outcome: Percentage of the Usage of Emergency Drugs
Time Frame: at the 4th week of follow-up
Population: ITT analysis was used
Measure: Number; unit: percentage of participants
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
percentage of participants | 10.53 | 12.50 | 30.43
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Deep Needling Group vs Shallow Needling Group; Test type: Superiority or Other; p = 0.587, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)
Statistical Analysis 3: Comparison: Deep Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.001, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)
Statistical Analysis 4: Comparison: Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p < 0.001, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)

10. Secondary Outcome: Percentage of the Usage of Emergency Drugs
Time Frame: at the 12th week of follow-up
Population: ITT analysis was used.
Measure: Number; unit: percentage of participants
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Number analyzed (Participants) | 228 | 112 | 115
percentage of participants | 17.11 | 14.29 | 29.57
Statistical Analysis 1: Comparison: Deep Needling Group vs Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.006, Chi-squared
Statistical Analysis 2: Comparison: Deep Needling Group vs Shallow Needling Group; Test type: Superiority or Other; p = 0.507, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)
Statistical Analysis 3: Comparison: Deep Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.005, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)
Statistical Analysis 4: Comparison: Shallow Needling Group vs Lactulose Group; Test type: Superiority or Other; p = 0.008, Chi-squared — α was corrected by the method of Bonferroni as 0.0167 (α=0.05/3=0.0167)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected in about more than two years.
Arm/Group | Deep Needling Group | Shallow Needling Group | Lactulose Group
Serious Adverse Events (participants affected / at risk) | 0/228 | 0/112 | 0/115
Other Adverse Events (participants affected / at risk) | 6/228 | 5/112 | 10/115
OTHER ADVERSE EVENTS (reported when occurring in more than 0.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Needling Group (N=228) | Shallow Needling Group (N=112) | Lactulose Group (N=115)
moderate or above pricking (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) — feelings of moderate or above pricking during the performance of needling
Subcutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) — Disappear in about 2 weeks
mild fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) — recover in 24 hours
diarrhea and abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 10 (10)

LIMITATIONS AND CAVEATS:
Spontaneous bowel movements were used as the primary outcome in our trial rather than complete, spontaneous bowel movements. Outcomes of follow-up were not the mean value of weekly data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes